CLINICAL TRIAL: NCT02062125
Title: A Prospective, Observational Study of Calcinosis in a Single-Center Population With Scleroderma-Spectrum Disorders
Brief Title: Calcinosis in a Single-Center Scleroderma Population
Acronym: SSc-calcinosis
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Vivien Hsu, M.D., Professor of Medicine, Rutgers, The State University of New Jersey
Other Study IDs: Pro2012001886
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Scleroderma; Calcinosis
Keywords: scleroderma; calcinosis
MeSH Terms: conditions — Scleroderma, Diffuse; Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a 10 year study of scleroderma patients with calcinosis 1) to better understand how common and if there are any risk factors for having calcinosis

2) to identify common complications associated with scleroderma-related calcinosis.

.

DETAILED DESCRIPTION:
This is a prospective study of scleroderma- spectrum patients focused on soft tissue calcinosis in order 1) to better understand the risk factors (including clinical/laboratory characteristics, and serology) of calcinosis in the scleroderma-spectrum disorders (limited or diffuse systemic sclerosis with or without overlap of inflammatory arthritis and/or myositis).

2) view common complications associated with calcinosis.

Better understanding of scleroderma calcinosis would lead to other studies that eventually will define better treatment options for this incurable and often disabling complication.

ELIGIBILITY:
Inclusion Criteria:

* Adult scleroderma subjects with and without calcinosis

Exclusion Criteria:

* Subjects unwilling to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult scleroderma subjects with and without calcinosis will be enrolled
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
risk factors and outcomes in scleroderma calcinosis | 10 years
  This is an observational study of scleroderma calcinosis to assess possible risk factors (including serologic studies and disease types) as well as common complications that occur in those with scleroderma calcinosis during this time period. We will assess for increased burden of calcinosis with associated musculoskeletal complications from calcinosis over 10 years.
  No additional intervention will be delivered, other than standard of care for this complication.

CONTACTS AND LOCATIONS:
Locations (1):
- RWJ Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No